CLINICAL TRIAL: NCT04813718
Title: Post COVID-19 Syndrome: A Pilot Study to Explore the Gut-lung Axis
Brief Title: Post COVID-19 Syndrome and the Gut-lung Axis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: CBmed Ges.m.b.H. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: PostCov
Record Dates: First submitted 2021-03-15; First posted 2021-03-24 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synbiotic (Active Comparator): Omni-Biotic Pro Vi 5
  Interventions: Dietary Supplement: Omni-Biotic Pro Vi 5
- Placebo (Placebo Comparator): similar looking and tasting
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omni-Biotic Pro Vi 5 — Pre- and probiotic
  Arms: Synbiotic
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The outbreak of the novel coronavirus (SARS-CoV-2)-infected disease (COVID-19) began in December 2019, spread throughout China in early 2020 and developed as a pandemic thereafter.

Based on current knowledge, Covid-19 infection causes mild to moderate respiratory and gastrointestinal symptoms in the majority of patients. In a smaller percentage severe disease courses are observed, often with the need of hospitalization and intensive care treatment. Apparently, symptoms can persist for relatively long time after viral clearance, suggesting the existence of a "Post-Covid" syndrome. A study from the UK identified fatigue, breathlessness and psychosocial stress as common symptoms after discharge from the hospital. Covid-19 infection is frequently characterized by a hyperinflammatory phenotype and a cytokine storm. The Covid-19 cytokine storm is characterised by rapid proliferation and hyperactivation of T cells, macrophages, mast cells, neutrophil granulocytes and natural killer cells, and the overproduction of inflammatory cytokines and chemical mediators released by immune or nonimmune cells. Early data also suggest that even if symptoms are just 'mild to moderate' during the acute infection, fibrotic lung damage develops in some patients. This may lead to long-term pulmonary complications for a subset of patients. The mechanisms for post-Covid pulmonary fibrosis are still unclear: inflammation triggering fibrosis, epithelial and endothelial injury with inadequate fibroproliferation and vascular damage are considered to be possible mechanisms.

A potential therapeutic target in ameliorating post-Covid symptoms could be the gut microbiome. Gut microbiome alterations have been described in Covid-19. The gut-lung axis as a link between dysbiosis, barrier dysfunction, translocation of bacterial products and hyperinflammation has been proposed as a potential therapeutic target. Probiotics have been proposed to be a possible modulator of the deranged gut-lung axis in Covid-disease and post-Covid syndrome. Currently 11 studies are registered in clinicaltrials.gov for treatment of acute Covid disease and prevention of the disease (including one study from Graz), but no study related to post-Covid syndrome could be found.

Therefore, it is currently unclear, which clinical, immune system or microbiome related biomarker would be the best to study the effect of a microbiome-based intervention in post-Covid syndrome.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Covid-19 infection with severe disease defined within the last 12 months (defined as one or more of the following: hospitalization, need for oxygen supply, need for intensive care treatment, need for specific treatment of Covid disease, antibiotic treatment)
* Subjective presence of residual symptoms of Covid disease OR no residual symptoms of Covid disease (Controls)
* Informed consent

Exclusion Criteria:

* Continuous probiotic treatment in the last 4 weeks before inclusion
* Pre-existing lung diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Microbiome composition | 6 months
  16 sRNA sequencing
Intestinal barrier | 6 months
  Change in zonulin levels over time and with/without the intervention
sCD14 | 6 months
  Change in sCD14 levels over time and with/without the intervention
endotoxin | 6 months
  Change in endotoxin levels serum over time and with/without the intervention
TNFalpha | 6 months
  Change in TNFalpha levels serum over time and with/without the intervention
Interleukin 1b | 6 months
  Change in Interleukin 1b serum levels over time and with/without the intervention
Interleukin 6 | 6 months
  Change in interleukin 6 serum levels over time and with/without the intervention
Interleukin 6 receptor | 6 months
  Change in Interleukin 6 receptor serum levels over time and with/without the intervention
interleukin 8 | 6 months
  Change in interleukin 8 serum levels over time and with/without the intervention
interleukin 10 | 6 months
  Change in interleukin 10 serum levels over time and with/without the intervention
interleukin 17 | 6 months
  Change in interleukin 17 serum levels over time and with/without the intervention
interleukin 23 | 6 months
  Change in interleukin 23 serum levels over time and with/without the intervention
neutrophil function burst function | 6 months
  Change in neutrophil burst function over time and with/without the intervention
neutrophil function phagocytosis | 6 months
  Change in neutrophil phagocytosis function over time and with/without the intervention
neutrophil NET formation | 6 months
  Change in neutrophil NET formation over time and with/without the intervention
neutrophil surface receptor expression | 6 months
  Change in neutrophil surface receptor expression over time and with/without the intervention
monocyte burst | 6 months
  Change in monocyte burst over time and with/without the intervention
monocyte phagocytosis | 6 months
  Change in monocyte phagocytosis over time and with/without the intervention
monocyte function surface receptor expression | 6 months
  Change in monocyte surface receptor expression over time and with/without the intervention
T cell immunophenotyping | 6 months
  Change in T cell subtypes over time and with/without the intervention
B cells immunophenotyping | 6 months
  Change in B cell subtypes over time and with/without the intervention
Spirometry | 6 months
  Change in spirometry measurements over time and with/without the intervention
Lung volume | 6 months
  Change in lung volume over time and with/without the intervention
Gas diffusion | 6 months
  Change in pulmonary gas diffusion over time and with/without the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No
Data will be shared upon reasonable request